CLINICAL TRIAL: NCT05313997
Title: The Incidence of Thoracic Disc Herniation in Patients Presenting With Chronic Upper Back Pain, A Follow-Up Study
Brief Title: The Incidence of Thoracic Disc Herniation in Patients Presenting With Chronic Upper Back Pain
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Emine Dundar Ahi, MD, Principal Investigator, Kocaeli University
Other Study IDs: 2022-20
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Thoracic Disc Herniation
Keywords: chronic upper back pain; thoracic disc herniation
MeSH Terms: interventions — Diclofenac; Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Diclofenac Sodium — at first diclofenac sodium was prescribed to patients with chronic upper back pain.
  If the patient's pain persisted, she/he was included in the physical therapy (hotpack 20 minutes, ultrason 5 minutes, Transcutaneous electrical nerve stimulation 20 minutes) program.
  Other Names: physical therapy

SUMMARY:
Patients who applied to the Private Medar Hospital between February 2016 and February 2021 with chronic upper back pain and were diagnosed with Thoaracic Disc Herniatin (TDH) (with Thoracic vertebral MRI) and followed up for at least 1 year will be included in the study.

Patients diagnosed with TDH were included in the medical treatment and/or physical therapy program.

Before and after these treatment programs, the pain intensity of the patients was recorded with the visual analog scale (VAS).

The number of patients who applied to the Physical Medicine and Rehabilitation outpatient clinic with chronic upper back pain between February 2016 and February 2021 will be researched, and the demographic characteristics of those diagnosed with TDH will be selected and recorded in their files, their pre- and post-treatment VAS scores, and the results will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* admitted to the Private Medar Hospital Gölcük hospital between February 2016 and February 2021 with chronic upper back pain.
* Diagnosed with TDH as a result of thoracic vertebral MRI

Exclusion Criteria:Patients with

* vertebral fracture,
* developmental spinal deformity,
* spinal infection or tumor,
* chronic widespread pain syndrome such as fibromyalgia,
* diabetes mellitus,
* polyneuropathy
* rheumatological disease
* under 18 years old
* over 65 years old
* who have had previous back and neck surgery

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * 18-65 years old
  * admitted to the Private Medar Hospital Gölcük hospital between February 2016 and February 2021 with chronic upper back pain.
  * Diagnosed with TDH as a result of thoracic vertebral MRI
Sampling Method: Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 10 seconds
  The Visual Analog Scale (VAS) is usually a 100-mm long horizontal line with verbal descriptors (word anchors) at each end to express the extremes of the feeling. FM patients mark the point on the line that best corresponds to their symptom severity. To this end, they are instructed to put a cross on the straight line at the point that most accurately expresses their degree of agreement. When reading the VAS, the position of the respondent's cross is generally assigned a score between 0 and 100. If documented in paper form, the scores can then be simply transferred to a 100- value scale using a millimeter tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: emine dundar ahi, ass professor, Principal Investigator — Kocaeli University
Locations (1):
- Private Medar Hospital, Kocaeli, Turkey (Türkiye)